CLINICAL TRIAL: NCT01834326
Title: A Randomized, Parallel-group Autogenous ex Vivo Produced Oral Mucosa Equivalent vs. Palatal Oral Mucosa Safety and Efficacy Study in Subjects Requiring Additional Keratinized Oral Mucosa for Dental Implants
Brief Title: Phase II Clinical Trial of Intraoral Grafting of Human Tissue Engineered Oral Mucosa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding period for the study ended. The study did not reach full enrollment.
Sponsor: Stephen E. Feinberg (Other)
Responsible Party: Sponsor-Investigator, Stephen E. Feinberg, Professor & Associate Chair of Research, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00065554
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Disorder of Oral Mucous Membrane
Keywords: dental implants; deficient keratinized oral mucosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palatal Oral Mucosa (POM) Graft (Active Comparator): Standard of care palatal oral mucosa (POM) graft will be taken from the palate and then surgically placed onto the defect area
  Interventions: Biological: POM (Palatal oral mucosa)
- Ex vivo Produced Oral Mucosa Equivalent (Experimental): Palatal biopsy will be harvested for fabrication of autogenous ex vivo produced oral mucosa equivalent (EVPOME) and then surgically placed onto the defect area
  Interventions: Biological: EVPOME (autogenous ex vivo produced oral mucosa equivalent)

INTERVENTIONS:
Biological: EVPOME (autogenous ex vivo produced oral mucosa equivalent) — EVPOME is manufactured from the subjects own oral cells and is implanted back in the subjects mouth after an approximately 30 day manufacturing process.
  Arms: Ex vivo Produced Oral Mucosa Equivalent
Biological: POM (Palatal oral mucosa) — POM is a tissue graft harvested from the palate and surgically placed into the defect area
  Arms: Palatal Oral Mucosa (POM) Graft

SUMMARY:
The purpose of this study is to improve the current standard of care of repairing mouth soft tissue defects.

DETAILED DESCRIPTION:
This study will test a tissue equivalent ex vivo produced oral mucosa equivalent(EVPOME), which is a subject's own cells grown on top of a piece of AlloDerm (a commercially available freeze dried human cadaver tissue that is routinely used in present day surgical reconstructive procedures) to create a new piece of soft tissue for use only in that subject's body. The tissue equivalent product will be tested against a non-experimental method of grafts, the gold standard a piece of palatal oral mucosa (POM) to see which works best. Each subject will be randomly assigned to receive either the EVPOME or POM to cover the defect in their mouth. The objective of the study is to assess the safety and efficacy for the use of human EVPOME for soft tissue intraoral grafting procedures compared to the "gold standard" palatal oral mucosa (POM) graft.

ELIGIBILITY:
Inclusion Criteria:

* Deficient band (<3mm) of keratinized mucosa prior to or following dental implant placement
* Surgery to increase width of keratinized mucosa is clinically indicated or requested by the patient to facilitate oral hygiene procedures or to improve esthetics
* Patients in need of a graft of approximately 15 x 10 x 20 mm in dimension

Exclusion Criteria:

* Subjects with potential medical complications such as evidence of clinically significant (as described by investigators) renal, hepatic, cardiac, endocrine, hematologic, autoimmune, or any systemic disease which may complication execution of the protocol and/or interpretation of results
* Current radiation therapy or history of radiation therapy treatment to the intraoral donor biopsy site or recipient site for graft placement
* Documented history of syphilis, HIV, Hepatitis B or C virus
* Pregnant women or women planning to become pregnant or unwilling to abstain or use double barrier contraceptives during the course of the study
* Smoking or use of tobacco products within 6 months prior to screening
* History of either alcohol or drug abuse
* Subjects taking medications that can result in gingival enlargement/overgrowth (Cyclosporine, Dilantin, calcium channel blockers)
* Current use of intravenous bisphosphonate or current oral bisphosphate use or a history of bisphosphonate use for over 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Feinberg, DDS, PhD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Department of Oral & Maxxillofacial Surgery, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent
Started | 10 | 8
Completed | 8 | 2
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Population: Surgery to increase width of keratinized mucosa is clinically indicated or requested by the patient to facilitate oral hygiene procedures or to improve esthetics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Customized [Count of Participants; unit: Participants]
  Age 18 to 80 Years | 10 | 8 | 18
Sex/Gender, Customized [Number; unit: participants]
  Male | 4 | 1 | 5
  Female | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 3 | 0 | 3
Deficient band of keratinized mucosa [Count of Participants; unit: Participants] — Patients referred to clinic requiring surgery to increase width of keratinized mucosa as clinically indicated or requested by the patient to facilitate oral hygiene procedures or to improve esthetics were eligible to consent for a study screening visit.
  Participants | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Clinical Increase in Zone (Width) of Keratinized Mucosa at Grafted Site
Description: The keratinized mucosa (KM) width will be measured by determining the distance from the crest of the edentulous ridge to the mucogingival line to the nearest millimeter with a Castroviejo caliper. The keratinized mucosa width of study subjects was measured prior to graft placement and then after two weeks, and after 4 weeks. The data provided shows the difference in keratinized mucosa width between the pre surgery measure and the post surgery measure. More mucosa width (positive numbers in mm) is an improvement, negative numbers (a decrease) would be less good.
Time Frame: 2 and 4 weeks post surgical graft
Population: Pregraft data for this outcome was not collected for the first subject, the protocol was written to collect the pregraft measurement after the first subject completed POM graft. For this reason there are only 7 data points in the POM arm of the study.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent
Number analyzed (Participants) | 7 | 2
millimeters
  2 Week increase in keratinized mucosa | 6.1 (1.9) | 6.5 (2.1)
  4 week increase in keratinized mucosa | 5.1 (1.4) | 4.5 (2.1)

2. Secondary Outcome: Graft Contracture
Description: Graft measurements collected at each time point post graft surgery, 2 weeks, 4 weeks, 8 weeks and 24 weeks. Measurements collected, Horizontal Coronal (mm), Horizontal Apical (mm), Vertical between coronal and apical (mm), were used to determine the area of the graft as a trapezoid like shape. The area of the graft at each time point was compared to the area of the graft at the time of implantation (graft surgery) to determine the % of graft contracture from implantation thru each follow-up time point. Less graft contracture is considered a better outcome.
Time Frame: 2, 4, 8 and 24 weeks after surgery
Measure: Mean (Standard Deviation); unit: Percentage of graft contracture
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent
Number analyzed (Participants) | 8 | 2
Percentage of graft contracture
  2 weeks post surgery | 10 (28) | 24 (34)
  4 weeks post surgery | 31 (24) | 49 (13)
  8 weeks post surgery | 45 (11) | 73 (4)
  24 weeks post surgery | 42 (15) | 71 (6)

3. Other Pre Specified Outcome: Graft Blood Flow
Description: Graft blood flow measured using Laser Doppler flowmetry (LDF) of the graft at 2 and 4 weeks after surgery. LDF measurements (perfusion units) are taken at the site of the graft and compared to LDF readings at a contralateral site on the same subject. The comparison is reported as a percent. The percent is derived by dividing the LDF perfusion units at the graft site by the LDF perfusion units at the contralateral site in the same subject. It is not known how many perfusion units are necessary to adequately supply blood to a graft. By comparing the graft site to the contralateral site in the same patient at 2 and 4 weeks post surgery this data may provide more understanding of graft incorporation.
Time Frame: 2 and 4 weeks after surgery
Measure: Mean (Standard Deviation); unit: Percent perfusion units graft/contralat
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent
Number analyzed (Participants) | 8 | 2
Percent perfusion units graft/contralat
  2 Week post surgery percent of perfusion units at graft site vs contralateral site on same subject | 202 (391) | 30 (4)
  4 week post surgery percent of perfusion units at graft site vs contralateral site on same subject | 206 (234) | 222 (210)

4. Other Pre Specified Outcome: Immunohistochemistry Using Anti-CD31 (Cluster of Differentiation 31) to Detect Blood Vessel Growth Into the Graft.
Description: A biopsy of the graft is taken at 4 weeks after engraftment. The biopsy is stained for CD31 (cluster of differentiation 31) which is a marker for blood vessels. The number of blood vessels are counted in a standardized size of field. The number of blood vessels within the standardized field is reported. It is not known how much blood vessel development is necessary for graft success, but this study may provide insight into blood vessel development within EVPOME grafts over time.
Time Frame: 4 weeks after graft surgery
Measure: Mean (Standard Deviation); unit: Number of blood vessels
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent
Number analyzed (Participants) | 8 | 2
Number of blood vessels | 15 (5) | 17 (7)

ADVERSE EVENTS:
Time Frame: Life of study, 3 years.
Arm/Group | Palatal Oral Mucosa (POM) Graft | Ex Vivo Produced Oral Mucosa Equivalent
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 6/10 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palatal Oral Mucosa (POM) Graft (N=10) | Ex Vivo Produced Oral Mucosa Equivalent (N=8)
Viral cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Temporary numbness in throat due to anesthetic (General disorders) | 1 (1) | 1 (1)
Herpes Labialis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Severed Tendon Right Bicep (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising, neck (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Throbbing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Keratin nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — 1 mm punctate ulceration noted with small hard 'keratin'" nodule in buccal mucosa
Stomach flu (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra oral herpes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lack of energy with feeling of fever (General disorders) | 1 (1) | 0 (0) — Lack of energy with feeling of fever.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT01834326/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT01834326/ICF_001.pdf